CLINICAL TRIAL: NCT04323124
Title: A PHASE 1, RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED, SINGLE AND MULTIPLE DOSE ESCALATION STUDY TO EVALUATE SAFETY, TOLERABILITY, PHARMACOKINETICS AND PHARMACODYNAMICS OF PF-07059013 AND OPEN-LABEL ASSESSMENT OF FOOD AND FORMULATION ON PHARMACOKINETICS OF PF-07059013 IN HEALTHY ADULT PARTICIPANTS
Brief Title: Study of Single and Multiple Ascending Doses of PF-07059013 in Healthy Adult Participants
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study was terminated as it did not demonstrate sufficient pharmacological effect. Termination was not related to safety reasons.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: C4061001; 2019-004918-34 (EudraCT Number)
Record Dates: First submitted 2020-03-18; First posted 2020-03-26 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-05

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): PF-07059013 assignment
  Interventions: Drug: PF-07059013
- Placebo (Placebo Comparator): Placebo assignment
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PF-07059013 — Participants will recieve PF-07059013
  Arms: Treatment
Drug: Placebo — Participants will recieve placebo
  Arms: Placebo

SUMMARY:
The purpose of the study is to evaluate the safety, tolerability, pharmacokinetics (PK) and pharmacodynamic (PD) of single and multiple ascending oral doses of PF-07059013 in healthy adult participants. Additionally, effects of different formulations and food on parameters, including PK may be explored.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female (of non-child bearing potential) participants must be 18 to 55 years of age, inclusive, at the time of signing the ICD.
2. Male and female participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, including blood pressure, pulse rate, respiratory rate and temperature measurement, standard 12 lead ECG, laboratory tests, and cardiac monitoring (in Part 1 only).
3. Participants who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures.

   Weight:
4. BMI of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lb).
5. Capable of giving signed informed consent as described in Appendix 1, which includes compliance with the requirements and restrictions listed in the ICD and in this protocol.

Exclusion Criteria

1. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
2. Any condition possibly affecting drug absorption (eg, gastrectomy, cholecystectomy).
3. History of human immunodeficiency virus (HIV) infection, hepatitis B, or hepatitis C; positive testing at screening for HIV, hepatitis B surface antigen (HBsAg), hepatitis B core antibody (HBcAb), or hepatitis C antibody (HCVAb). As an exception a positive HBsAb test due to hepatitis B vaccination is permissible.
4. Other medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
5. Use of prescription or nonprescription drugs and dietary and herbal supplements within 7 days or 5 half lives (whichever is longer) prior to the first dose of study intervention.
6. Previous administration with an investigational drug within 30 days (or as determined by the local requirement) or 5 half lives preceding the first dose of study intervention used in this study (whichever is longer).
7. A positive urine drug test at screening or admission.
8. A positive urine cotinine test at screening or admission in Part 1 and 2.
9. Screening supine BP ≥140 mm Hg (systolic) or ≥90 mm Hg (diastolic), following at least 5 minutes of supine rest. If BP is ≥140 mm Hg (systolic) or ≥90 mm Hg (diastolic), the BP should be repeated 2 more times and the average of the 3 BP values should be used to determine the participant's eligibility.
10. Baseline 12 lead ECG that demonstrates clinically relevant abnormalities that may affect participant safety or interpretation of study results (eg, baseline QTc interval >450 msec, complete left bundle branch block (LBBB), signs of an acute or indeterminate age myocardial infarction, ST T interval changes suggestive of myocardial ischemia, second or third degree atrioventricular (AV) block, or serious bradyarrhythmias or tachyarrhythmias). If the baseline uncorrected QT interval is >450 msec, this interval should be rate corrected using the Fridericia method and the resulting QTcF should be used for decision making and reporting. If QTc exceeds 450 msec, or QRS exceeds 120 msec, the ECG should be repeated 2 more times and the average of the 3 QTc or QRS values should be used to determine the participant's eligibility. Computer interpreted ECGs should be overread by a physician experienced in reading ECGs before excluding participants.
11. Participants with ANY of the following abnormalities in clinical laboratory tests at screening, as assessed by the study specific laboratory and confirmed by a single repeat test, if deemed necessary:

    * AST or ALT level ≥1.5 × ULN;
    * Total bilirubin level ≥1.5 × ULN; participants with a history of Gilbert's syndrome may have direct bilirubin measured and would be eligible for this study provided the direct bilirubin level is ≤ ULN;
    * PT/INR >1.2 × ULN;
    * aPTT ≥1.5 × ULN;
    * Hemoglobin <11.0 g/dL;
    * Lactate >1 x ULN.
12. For Part 2 only, participants with absolute reticulocyte count >150,000/uL at screening, as assessed by the study specific laboratory and confirmed by a single repeat test, if deemed necessary.
13. History of alcohol abuse or binge drinking and/or any other illicit drug use or dependence within 6 months of Screening. Binge drinking is defined as a pattern of 5 (male) and 4 (female) or more alcoholic drinks in about 2 hours. As a general rule, alcohol intake should not exceed 14 units per week (1 unit = 8 ounces (240 mL) beer, 1 ounce (30 mL) of 40% spirit or 3 ounces (90 mL) of wine).
14. Use of tobacco/nicotine containing products for Part 1 or 2, and use of more than 5 cigarettes/day for Part 3.
15. Blood donation (excluding plasma donations) of approximately 1 pint (500 mL) or more within 60 days prior to dosing.
16. Unwilling or unable to comply with the criteria in the Lifestyle Considerations section of this protocol.
17. Investigator site staff or Pfizer employees directly involved in the conduct of the study, site staff otherwise supervised by the investigator, and their respective family members.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2020-07-17 (Actual); Primary Completion 2021-10-21 (Actual); Study Completion 2021-10-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Clinical Research Unit - Brussels, Brussels, Bruxelles-capitale, Région de, Belgium

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Lee KC, Wan KX, Barricklow J, Lim CN, Clarke S, Potts D, Holmes K, Gonzalez P, Kavetska O. Using Mitra sampling to support first-in-human pharmacokinetic evaluations for PF-07059013. Bioanalysis. 2023 Sep;15(17):1083-1094. doi: 10.4155/bio-2023-0066. Epub 2023 Aug 16. PMID 37584365
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4061001

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 61 participants were randomized in the study and all were treated with study intervention.
  For Part 1, a total of 21 participants were randomized and all were treated with at least 1 dose.
  For Part 2, a total of 35 participants were randomized and treated.
  For Part 3, a total of 5 participants were randomized and all were treated with at least 1 dose.
Groups:
- A->D->F->H: In Part 1, participants were given a single dose of each study intervention assigned.
  A->D->F->H: Placebo Single dose (SD) Polymer->PF-07059013 500 mg SD Polymer->PF-07059013 2000 mg SD Polymer->PF-07059013 2000 mg SD without (w/o) Polymer
- A->E->G->I: In Part 1, participants were given a single dose of each study intervention assigned.
  A->E->G->I: Placebo SD Polymer->PF-07059013 1000 mg SD Polymer->PF-07059013 3000 mg SD Polymer->PF-07059013 3000 mg SD w/o Polymer
- B->A->F->H: In Part 1, participants were given a single dose of each study intervention assigned.
  B->A->F->H: PF-07059013 100 mg SD Polymer->Placebo SD Polymer->PF-07059013 2000 mg SD Polymer->PF-07059013 2000 mg SD w/o Polymer
- B->D->A->H: In Part 1, participants were given a single dose of each study intervention assigned.
  B->D->A->H: PF-07059013 100 mg SD Polymer->PF-07059013 500 mg SD Polymer->Placebo SD Polymer->PF-07059013 2000 mg SD w/o Polymer
- C->A->G->I: In Part 1, participants were given a single dose of each study intervention assigned.
  C->A->G->I: PF-07059013 250 mg SD Polymer->Placebo SD Polymer->PF-07059013 3000 mg SD Polymer->PF-07059013 3000 mg SD w/o Polymer
- C->E->A->I: In Part 1, participants were given a single dose of each study intervention assigned.
  C->E->A->I: PF-07059013 250 mg SD Polymer->PF-07059013 1000 mg SD Polymer->Placebo SD Polymer->PF-07059013 3000 mg SD w/o Polymer
- Placebo MD; PF-07059013 800 mg MD; PF-07059013 1600 mg MD; PF-07059013 3000 mg MD; PF-07059013 4000 mg MD: In Part 2, participants were given multiple doses of study intervention once daily (QD) for 14 days.
- P->Q->R->S: In Part 3, participants were given a single dose of study intervention assigned under fasted conditions. The presence/absence of polymer is utilized to select the preferred formulation composition.
  P->Q->R->S:Suspension Fasted Polymer (Small Particle Size)->Tablet Fasted w/o Polymer->Suspension Fed Polymer (Small Particle Size)->Suspension Fasted Polymer (Moderate Particle Size)
- P->Q->S->R: In Part 3, participants were given a single dose of study intervention assigned under fasted conditions. The presence/absence of polymer is utilized to select the preferred formulation composition.
  P->Q->S->R: Suspension Fasted Polymer (Small Particle Size)->Tablet Fasted w/o Polymer->Suspension Fasted Polymer (Moderate Particle Size)->Suspension Fed Polymer (Small Particle Size)
- Q->P->R->S: In Part 3, participants were given a single dose of study intervention assigned under fasted conditions. The presence/absence of polymer is utilized to select the preferred formulation composition.
  Q->P->R->S: Tablet Fasted w/o Polymer->Suspension Fasted Polymer (Small Particle Size)->Suspension Fed Polymer (Small Particle Size)->Suspension Fasted Polymer (Moderate Particle Size)
- Q->P->S->R: In Part 3, participants were given a single dose of study intervention assigned under fasted conditions. The presence/absence of polymer is utilized to select the preferred formulation composition.
  Q->P->S->R: Tablet Fasted w/o Polymer->Suspension Fasted Polymer (Small Particle Size)->Suspension Fasted Polymer (Moderate Particle Size)->Suspension Fed Polymer (Small Particle Size)
Period: Overall Study
Arm/Group | A->D->F->H | A->E->G->I | B->A->F->H | B->D->A->H | C->A->G->I | C->E->A->I | Placebo MD | PF-07059013 800 mg MD | PF-07059013 1600 mg MD | PF-07059013 3000 mg MD | PF-07059013 4000 mg MD | P->Q->R->S | P->Q->S->R | Q->P->R->S | Q->P->S->R
Started | 3 | 3 | 3 | 3 | 5 | 4 | 8 | 8 | 7 | 6 | 6 | 2 | 1 | 1 | 1
Completed | 3 | 3 | 3 | 3 | 3 | 2 | 8 | 6 | 5 | 6 | 6 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 2 | 2 | 0 | 0 | 2 | 1 | 1 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Coming from a red zone (COVID) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — No longer meets eligibility criteria | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Study terminated by sponsor | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- A->D->F->H: In Part 1, participants were given a single dose of study intervention assigned.
  A->D->F->H: Placebo Single dose (SD) Polymer->PF-07059013 500 mg SD Polymer->PF-07059013 2000 mg SD Polymer->PF-07059013 2000 mg SD without (w/o) Polymer
- A->E->G->I: In Part 1, participants were given a single dose of study intervention assigned.
  A->E->G->I: Placebo SD Polymer->PF-07059013 1000 mg SD Polymer->PF-07059013 3000 mg SD Polymer->PF-07059013 3000 mg SD w/o Polymer
- B->A->F->H: In Part 1, participants were given a single dose of study intervention assigned.
  B->A->F->H: PF-07059013 100 mg SD Polymer->Placebo SD Polymer->PF-07059013 2000 mg SD Polymer->PF-07059013 2000 mg SD w/o Polymer
- B->D->A->H: In Part 1, participants were given a single dose of study intervention assigned.
  B->D->A->H: PF-07059013 100 mg SD Polymer->PF-07059013 500 mg SD Polymer->Placebo SD Polymer->PF-07059013 2000 mg SD w/o Polymer
- C->A->G->I: In Part 1, participants were given a single dose of study intervention assigned.
  C->A->G->I: PF-07059013 250 mg SD Polymer->Placebo SD Polymer->PF-07059013 3000 mg SD Polymer->PF-07059013 3000 mg SD w/o Polymer
- C->E->A->I: In Part 1, participants were given a single dose of study intervention assigned.
  C->E->A->I: PF-07059013 250 mg SD Polymer->PF-07059013 1000 mg SD Polymer->Placebo SD Polymer->PF-07059013 3000 mg SD w/o Polymer
- Part 2: Placebo MD With Polymer; Part 2: PF-07059013 800 mg MD With Polymer; Part 2: PF-07059013 1600 mg MD With Polymer; Part 2: PF-07059013 3000 mg MD With Polymer; Part 2: PF-07059013 4000 mg MD With Polymer: In Part 2, participants were given multiple doses of study intervention QD for 14 days.
- P->Q->R->S: In Part 3, participants were given a single dose of study intervention assigned under fed or fasted conditions.
  P->Q->R->S: Suspension Fasted Polymer (Small Particle Size)->Tablet Fasted w/o Polymer->Suspension Fed Polymer (Small Particle Size)->Suspension Fasted Polymer (Moderate Particle Size)
- P->Q->S->R: In Part 3, participants were given a single dose of study intervention assigned under fed or fasted conditions.
  P->Q->S->R: Suspension Fasted Polymer (Small Particle Size)->Tablet Fasted w/o Polymer->Suspension Fasted Polymer (Moderate Particle Size)->Suspension Fed Polymer (Small Particle Size)
- Q->P->R->S: In Part 3, participants were given a single dose of study intervention assigned under fed or fasted conditions.
  Q->P->R->S: Tablet Fasted w/o Polymer->Suspension Fasted Polymer (Small Particle Size)->Suspension Fed Polymer (Small Particle Size)->Suspension Fasted Polymer (Moderate Particle Size)
- Q->P->S->R: In Part 3, participants were given a single dose of study intervention assigned under fed or fasted conditions.
  Q->P->S->R: Tablet Fasted w/o Polymer->Suspension Fasted Polymer (Small Particle Size)->Suspension Fasted Polymer (Moderate Particle Size)->Suspension Fed Polymer (Small Particle Size)
- Total: Total of all reporting groups
Arm/Group | A->D->F->H | A->E->G->I | B->A->F->H | B->D->A->H | C->A->G->I | C->E->A->I | Part 2: Placebo MD With Polymer | Part 2: PF-07059013 800 mg MD With Polymer | Part 2: PF-07059013 1600 mg MD With Polymer | Part 2: PF-07059013 3000 mg MD With Polymer | Part 2: PF-07059013 4000 mg MD With Polymer | P->Q->R->S | P->Q->S->R | Q->P->R->S | Q->P->S->R | Total
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 5 | 4 | 8 | 8 | 7 | 6 | 6 | 2 | 1 | 1 | 1 | 61
Age, Customized [Number; unit: Participants]
  <18 Years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  18-25 Years | 0 | 0 | 0 | 0 | 1 | 0 | 4 | 4 | 1 | 2 | 2 | 0 | 0 | 0 | 1 | 15
  26-35 Years | 0 | 1 | 1 | 1 | 2 | 1 | 1 | 2 | 4 | 3 | 2 | 0 | 0 | 0 | 0 | 18
  36-45 Years | 2 | 1 | 1 | 1 | 0 | 2 | 3 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 14
  >45 Years | 1 | 1 | 1 | 1 | 2 | 1 | 0 | 1 | 2 | 0 | 1 | 2 | 0 | 1 | 0 | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 3 | 3 | 3 | 3 | 5 | 4 | 8 | 8 | 7 | 6 | 6 | 2 | 1 | 1 | 1 | 61
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 3 | 3 | 3 | 3 | 5 | 2 | 7 | 7 | 5 | 5 | 6 | 2 | 1 | 1 | 1 | 54
  Black or African American | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 4
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Not reported | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Race/Ethnicity, Customized [Number; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 1 | 3 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 9
  Not Hispanic or Latino | 2 | 3 | 3 | 2 | 2 | 3 | 8 | 7 | 6 | 6 | 5 | 2 | 1 | 1 | 1 | 52

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Treatment-Related Adverse Event(s) (Treatment-Related TEAE)
Description: Adverse events (AEs): any untoward medical occurrence in a clinical investigation participant administered a product or medical device, without regard to causality. Treatment-emergent AEs (TEAEs): AEs which occurred for the first time during the effective duration of treatment or AEs that increased in severity during treatment. Treatment-related TEAEs were any untoward medical occurrence attributed to study intervention. Relatedness to study treatment was determined by the investigator.
  Duration of participation of Part 1 and Part 3, from the screening visit to the follow-up phone call, was approximately 15 weeks. Duration of participation of Part 2, from the screening visit to the follow-up phone call, was approximately 10 weeks.
Time Frame: Baseline up to Follow-Up (15 weeks in Part 1 and Part 3, and 10 weeks in Part 2)
Population: All participants randomly assigned to study intervention and who took at least 1 dose of study intervention were included in safety analysis set. Participants were analyzed according to the product they actually received.
Measure: Count of Participants; unit: Participants
Groups:
- Part 1: Placebo Single Dose (SD) With Polymer: In Part 1, participants were given a single dose of study intervention assigned. The presence/absence of polymer is utilized to select the preferred formulation composition.
- Part 1: PF-07059013 100 mg SD With Polymer; Part 1: PF-07059013 250 mg SD With Polymer; Part 1: PF-07059013 500 mg SD With Polymer; Part 1: PF-07059013 1000 mg SD With Polymer; Part 1: PF-07059013 2000 mg SD With Polymer; Part 1: PF-07059013 3000 mg SD With Polymer; Part 1: PF- 07059013 2000 mg SD Without Polymer; Part 1: PF-07059013 3000 mg SD Without Polymer: In Part 1, participants were given a single dose of study intervention assigned.
- Part 2: Placebo Multiple Doses (MD) With Polymer: In Part 2, participants were given multiple doses of study intervention once daily (QD) for 14 days. The presence/absence of polymer is utilized to select the preferred formulation composition.
- Part 3: Suspension Fasted Polymer (Small Particle Size): In Part 3, participants were given a single dose of study intervention assigned under fasted conditions. The presence/absence of polymer is utilized to select the preferred formulation composition.
- Part 3: Tablet Fasted Without Polymer: In Part 3, participants were given a single dose of study intervention assigned under fasted conditions.
- Part 3: Suspension Fed Polymer (Small Particle Size): In Part 3, participants were given a single dose of study intervention assigned under fed conditions.
Arm/Group | Part 1: Placebo Single Dose (SD) With Polymer | Part 1: PF-07059013 100 mg SD With Polymer | Part 1: PF-07059013 250 mg SD With Polymer | Part 1: PF-07059013 500 mg SD With Polymer | Part 1: PF-07059013 1000 mg SD With Polymer | Part 1: PF-07059013 2000 mg SD With Polymer | Part 1: PF-07059013 3000 mg SD With Polymer | Part 1: PF- 07059013 2000 mg SD Without Polymer | Part 1: PF-07059013 3000 mg SD Without Polymer | Part 2: Placebo Multiple Doses (MD) With Polymer | Part 2: PF-07059013 800 mg MD With Polymer | Part 2: PF-07059013 1600 mg MD With Polymer | Part 2: PF-07059013 3000 mg MD With Polymer | Part 2: PF-07059013 4000 mg MD With Polymer | Part 3: Suspension Fasted Polymer (Small Particle Size) | Part 3: Tablet Fasted Without Polymer | Part 3: Suspension Fed Polymer (Small Particle Size)
Number analyzed (Participants) | 18 | 6 | 5 | 6 | 6 | 6 | 6 | 9 | 8 | 8 | 8 | 7 | 6 | 6 | 3 | 4 | 1
Participants
  All-causality | 3 | 2 | 2 | 0 | 1 | 0 | 4 | 2 | 4 | 4 | 7 | 7 | 4 | 5 | 3 | 2 | 0
  Treatment-related | 2 | 1 | 1 | 0 | 1 | 0 | 3 | 1 | 3 | 4 | 6 | 6 | 4 | 5 | 2 | 2 | 0

2. Primary Outcome: Number of Participants With Laboratory Test Findings of Potential Clinical Importance
Description: Protocol-required safety laboratory assessments included chemistry, hematology, and urinalysis (and microscopy, if needed). Each parameter was evaluated against commonly used and widely accepted criteria. Laboratory test with abnormalities are reported.
  Evaluation activities as:
  Part 1: At Screening, Day -1, and Day 1 (at 8 hours post dose), 2, 5, 8. Part 2: At Screening, Day -1, 1, 2, 4, 7, 10, 14, 18, 21. Part 3: At Screening, Day -1, 2, 5.
Time Frame: Part 1: from Screening to Day 8; Part 2: from Screening to Day 21; Part 3: from Screening to Day 5.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Part 2: Placebo Multiple Doses (MD) With Polymer: In Part 2, participants were given multiple doses of study intervention once daily (QD) for 14 days.
Arm/Group | Part 1: Placebo Single Dose (SD) With Polymer | Part 1: PF-07059013 100 mg SD With Polymer | Part 1: PF-07059013 250 mg SD With Polymer | Part 1: PF-07059013 500 mg SD With Polymer | Part 1: PF-07059013 1000 mg SD With Polymer | Part 1: PF-07059013 2000 mg SD With Polymer | Part 1: PF-07059013 3000 mg SD With Polymer | Part 1: PF- 07059013 2000 mg SD Without Polymer | Part 1: PF-07059013 3000 mg SD Without Polymer | Part 2: Placebo Multiple Doses (MD) With Polymer | Part 2: PF-07059013 800 mg MD With Polymer | Part 2: PF-07059013 1600 mg MD With Polymer | Part 2: PF-07059013 3000 mg MD With Polymer | Part 2: PF-07059013 4000 mg MD With Polymer | Part 3: Suspension Fasted Polymer (Small Particle Size) | Part 3: Tablet Fasted Without Polymer | Part 3: Suspension Fed Polymer (Small Particle Size)
Number analyzed (Participants) | 18 | 6 | 5 | 6 | 6 | 6 | 6 | 9 | 8 | 8 | 8 | 7 | 6 | 6 | 3 | 4 | 1
Participants
  Reticulocytes (10^9/L) >1.5 x upper limit of normal (ULN) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 1 | 2 | 0 | 0 | 0
  Reticulocytes/Erythrocytes (L/L) >1.5 x ULN | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0
  Lymphocytes/Leukocytes (%) <0.8 x lower limit of normal (LLN) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Neutrophils(10^9/L) <0.8 x LLN | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophils/Leukocytes (%) <0.8 x LLN | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Eosinophils (10^9/L) >1.2 x ULN | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Eosinophils/Leukocytes (%) >1.2 x ULN | 1 | 1 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
  Monocytes(10^9/L) >1.2 x ULN | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Monocytes/Leukocytes (%) >1.2 x ULN | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0
  Erythropoietin (IU/L) >1.0 x ULN | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Direct Bilirubin (micromol/L) >1.5 x ULN | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
  Urea Nitrogen (mmol/L) >1.3 x ULN | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Urea (mmol/L) >1.3 x ULN | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lactic Acid (mmol/L) >1.0 x ULN | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Specific Gravity (Urinalysis) <1.003 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
  URINE Bilirubin >=1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  URINE Protein >=1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  URINE Hemoglobin >=1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Leukocyte Esterase (Urinalysis) >=1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

3. Primary Outcome: Number of Participants With Vital Signs Findings of Potential Clinical Importance
Description: Vital sign data included supine blood pressure, pulse rate, orthostatic blood pressure and oral temperature. Vital signs with abnormalities are reported.
  Evaluation activities as:
  Part 1: Supine blood pressure and pulse rate: At Screening, 0, 0.5, 1, 2, 5, 8, 12, 24, 36, 48, 72, 96, and 168 hours post dose. Orthostatic blood pressure, respiratory rate and oral temperature: 0, 2, 8, and 24 hours post dose.
  Part 2: Supine blood pressure and pulse rate: At Screening, Day 1, 2, 4, 7, 10, 14, 15, 18, 21. Orthostatic blood pressure, respiratory rate and oral temperature: Day 1, 7, 14, 18.
  Part 3: Supine blood pressure and pulse rate: At Screening, 0, 2, 5, 8, 12, 24, 48, and 96 hours post dose. Respiratory rate and oral temperature: 0, 24 and 96 hours post dose.
Time Frame: Part 1: from Screening to Day 8; Part 2: from Screening to Day 21; Part 3: from Screening to Day 5.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Placebo Single Dose (SD) With Polymer | Part 1: PF-07059013 100 mg SD With Polymer | Part 1: PF-07059013 250 mg SD With Polymer | Part 1: PF-07059013 500 mg SD With Polymer | Part 1: PF-07059013 1000 mg SD With Polymer | Part 1: PF-07059013 2000 mg SD With Polymer | Part 1: PF-07059013 3000 mg SD With Polymer | Part 1: PF- 07059013 2000 mg SD Without Polymer | Part 1: PF-07059013 3000 mg SD Without Polymer | Part 2: Placebo Multiple Doses (MD) With Polymer | Part 2: PF-07059013 800 mg MD With Polymer | Part 2: PF-07059013 1600 mg MD With Polymer | Part 2: PF-07059013 3000 mg MD With Polymer | Part 2: PF-07059013 4000 mg MD With Polymer | Part 3: Suspension Fasted Polymer (Small Particle Size) | Part 3: Tablet Fasted Without Polymer | Part 3: Suspension Fed Polymer (Small Particle Size)
Number analyzed (Participants) | 18 | 6 | 5 | 6 | 6 | 6 | 6 | 9 | 8 | 8 | 8 | 7 | 6 | 6 | 3 | 4 | 1
Participants
  Supine Systolic Blood Pressure (mmHg) Value <90 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Supine Systolic Blood Pressure (mmHg) Change >=30 increase | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Supine Systolic Blood Pressure (mmHg) Change >=30 decrease | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Supine Diastolic Blood Pressure (mmHg) Value <50 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Supine Diastolic Blood Pressure (mmHg) Change >=20 increase | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Supine Diastolic Blood Pressure (mmHg) Change >=20 decrease | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Supine Pulse Rate (beats/min) Value <40 bpm | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Supine Pulse Rate (beats/min) Value >120 bpm | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Electrocardiogram (ECG) Findings of Potential Clinical Importance
Description: Clinical significance of 12-Lead ECG data was assessed by the investigator. ECG findings with abnormalities were reported.
  Evaluation activities as:
  Part 1: At Screening, 0, 0.5, 1, 2, 5, 8, 12, 24, 36, 48, 72, 96, and 168 hours post dose.
  Part 2: At Screening, Day 1, 2, 4, 7, 10, 14, 15, 18, 21. Part 3: At Screening, 0, 2, 5, 8, 12, 24, 48, and 96 hours post dose.
Time Frame: Part 1: from Screening to Day 8; Part 2: from Screening to Day 21; Part 3: from Screening to Day 5.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Placebo Single Dose (SD) With Polymer | Part 1: PF-07059013 100 mg SD With Polymer | Part 1: PF-07059013 250 mg SD With Polymer | Part 1: PF-07059013 500 mg SD With Polymer | Part 1: PF-07059013 1000 mg SD With Polymer | Part 1: PF-07059013 2000 mg SD With Polymer | Part 1: PF-07059013 3000 mg SD With Polymer | Part 1: PF- 07059013 2000 mg SD Without Polymer | Part 1: PF-07059013 3000 mg SD Without Polymer | Part 2: Placebo Multiple Doses (MD) With Polymer | Part 2: PF-07059013 800 mg MD With Polymer | Part 2: PF-07059013 1600 mg MD With Polymer | Part 2: PF-07059013 3000 mg MD With Polymer | Part 2: PF-07059013 4000 mg MD With Polymer | Part 3: Suspension Fasted Polymer (Small Particle Size) | Part 3: Tablet Fasted Without Polymer | Part 3: Suspension Fed Polymer (Small Particle Size)
Number analyzed (Participants) | 18 | 6 | 5 | 6 | 6 | 6 | 6 | 9 | 8 | 8 | 8 | 7 | 6 | 6 | 3 | 4 | 1
Participants
  PR Interval, Aggregate (msec) %Change>=25/50 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QTCB Interval, Aggregate (msec), 450<Value<480 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QTCB Interval, Aggregate (msec), 30<=Change<=60 | 2 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 4 | 1 | 0 | 1 | 2 | 0 | 0 | 0
  QTCF interval, Aggregate (msec), 30<=Change<=60 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: PF-07059013 Blood and Plasma Maximum Observed Concentration (Cmax) of Part 1
Description: PF-07059013 Blood and Plasma Cmax for Part 1 was evaluated. For Part 1, in period 1, participants were given PF-07059013 100 mg SD and PF-07059013 250 mg SD, all with polymer; in period 2, participants were given PF-07059013 500 mg SD and PF-07059013 1000 mg SD, all with polymer; in period 3, participants were given PF-07059013 2000 mg SD and PF-07059013 3000 mg SD, all with polymer; in period 4, participants were given PF-07059013 2000 mg SD and PF-07059013 3000 mg SD, all without polymer.
Time Frame: 0, 0.5, 1, 2, 5, 8, 12, 24, 36, 48, 72 (period 2-4 only), 96 (period 2-4 only), and 168 hours post dose of each period.
Population: The analysis population referred to all participants dosed who had at least 1 of the pharmacokinetics (PK) parameters of secondary interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Part 1: PF-07059013 100 mg SD With Polymer | Part 1: PF-07059013 250 mg SD With Polymer | Part 1: PF-07059013 500 mg SD With Polymer | Part 1: PF-07059013 1000 mg SD With Polymer | Part 1: PF-07059013 2000 mg SD With Polymer | Part 1: PF-07059013 3000 mg SD With Polymer | Part 1: PF- 07059013 2000 mg SD Without Polymer | Part 1: PF-07059013 3000 mg SD Without Polymer
Number analyzed (Participants) | 6 | 5 | 6 | 6 | 6 | 6 | 9 | 8
nanogram per milliliter (ng/mL)
  Blood | 4773 (36) | 11990 (43) | 25140 (51) | 52830 (38) | 104200 (63) | 231700 (31) | 107000 (54) | 191700 (55)
  Plasma | 88.51 (19) | 160.2 (31) | 250.1 (32) | 509.2 (22) | 555.3 (30) | 917.7 (38) | 496.1 (32) | 796.5 (39)

6. Secondary Outcome: PF-07059013 Blood and Plasma Time for Cmax (Tmax) of Part 1
Description: PF-07059013 Blood and Plasma Tmax for Part 1 was evaluated. For Part 1, in period 1, participants were given PF-07059013 100 mg SD and PF-07059013 250 mg SD, all with polymer; in period 2, participants were given PF-07059013 500 mg SD and PF-07059013 1000 mg SD, all with polymer; in period 3, participants were given PF-07059013 2000 mg SD and PF-07059013 3000 mg SD, all with polymer; in period 4, participants were given PF-07059013 2000 mg SD and PF-07059013 3000 mg SD, all without polymer.
Time Frame: 0, 0.5, 1, 2, 5, 8, 12, 24, 36, 48, 72 (period 2-4 only), 96 (period 2-4 only), and 168 hours post dose of each period.
Population: The analysis population referred to all participants dosed who had at least 1 of the PK parameters of secondary interest.
Measure: Median (Full Range); unit: hour
Arm/Group | Part 1: PF-07059013 100 mg SD With Polymer | Part 1: PF-07059013 250 mg SD With Polymer | Part 1: PF-07059013 500 mg SD With Polymer | Part 1: PF-07059013 1000 mg SD With Polymer | Part 1: PF-07059013 2000 mg SD With Polymer | Part 1: PF-07059013 3000 mg SD With Polymer | Part 1: PF- 07059013 2000 mg SD Without Polymer | Part 1: PF-07059013 3000 mg SD Without Polymer
Number analyzed (Participants) | 6 | 5 | 6 | 6 | 6 | 6 | 9 | 8
hour
  Blood | 1.00 [0.500 to 1.00] | 1.00 [0.500 to 1.00] | 1.00 [1.00 to 2.00] | 2.00 [1.00 to 2.07] | 2.00 [2.00 to 5.00] | 5.00 [2.00 to 5.00] | 2.03 [2.00 to 5.00] | 2.00 [2.00 to 5.00]
  Plasma | 1.00 [0.517 to 2.02] | 1.00 [0.500 to 2.00] | 2.00 [0.600 to 2.00] | 2.00 [1.00 to 8.00] | 2.00 [2.00 to 2.12] | 3.57 [2.00 to 5.00] | 2.03 [1.00 to 5.00] | 2.01 [2.00 to 8.00]

7. Secondary Outcome: PF-07059013 Blood and Plasma Area Under the Concentration-Time Profile From Time 0 to the Time of the Last Quantifiable Concentration (AUClast) of Part 1
Description: PF-07059013 Blood and Plasma AUClast of Part 1 was evaluated. For Part 1, in period 1, participants were given PF-07059013 100 mg SD and PF-07059013 250 mg SD, all with polymer; in period 2, participants were given PF-07059013 500 mg SD and PF-07059013 1000 mg SD, all with polymer; in period 3, participants were given PF-07059013 2000 mg SD and PF-07059013 3000 mg SD, all with polymer; in period 4, participants were given PF-07059013 2000 mg SD and PF-07059013 3000 mg SD, all without polymer.
Time Frame: 0, 0.5, 1, 2, 5, 8, 12, 24, 36, 48, 72 (period 2-4 only), 96 (period 2-4 only), and 168 hours post dose of each period.
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*hr/mL)
Arm/Group | Part 1: PF-07059013 100 mg SD With Polymer | Part 1: PF-07059013 250 mg SD With Polymer | Part 1: PF-07059013 500 mg SD With Polymer | Part 1: PF-07059013 1000 mg SD With Polymer | Part 1: PF-07059013 2000 mg SD With Polymer | Part 1: PF-07059013 3000 mg SD With Polymer | Part 1: PF- 07059013 2000 mg SD Without Polymer | Part 1: PF-07059013 3000 mg SD Without Polymer
Number analyzed (Participants) | 6 | 5 | 6 | 6 | 6 | 6 | 9 | 8
nanogram*hour per milliliter (ng*hr/mL)
  Blood | 14870 (49) | 73300 (45) | 211400 (65) | 639800 (47) | 1582000 (68) | 4091000 (34) | 1692000 (69) | 3562000 (77)
  Plasma | 520.5 (45) | 1699 (28) | 3224 (37) | 7505 (24) | 12310 (16) | 20520 (26) | 12640 (30) | 19130 (56)

8. Secondary Outcome: PF-07059013 Blood and Plasma Cmax of Part 2
Description: PF-07059013 Blood and Plasma Cmax of Part 2 was evaluated.
Time Frame: 0, 0.5, 1, 2, 4, 6, 8, 12 hours post dose on Day 1, 7, and 14.
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 2: PF-07059013 800 mg MD With Polymer | Part 2: PF-07059013 1600 mg MD With Polymer | Part 2: PF-07059013 3000 mg MD With Polymer | Part 2: PF-07059013 4000 mg MD With Polymer
Number analyzed (Participants) | 8 | 7 | 6 | 6
ng/mL
  Day 1 in Blood | 57230 (20) | 149500 (29) | 332100 (27) | 337500 (37)
  Day 1 in Plasma | 427.1 (23) | 597.2 (24) | 1071 (21) | 1339 (29)
  Day 7 in Blood: number analyzed (Participants) | 7 | 4 | 6 | 6
  Day 7 in Blood | 86020 (18) | 275700 (28) | 521600 (38) | 576900 (17)
  Day 7 in Plasma: number analyzed (Participants) | 7 | 4 | 6 | 6
  Day 7 in Plasma | 513.6 (22) | 913.9 (40) | 1496 (23) | 2157 (32)
  Day 14 in Blood: number analyzed (Participants) | 6 | 5 | 6 | 6
  Day 14 in Blood | 79690 (21) | 275800 (28) | 520000 (20) | 623700 (22)
  Day 14 in Plasma: number analyzed (Participants) | 6 | 5 | 6 | 6
  Day 14 in Plasma | 569.4 (44) | 868.2 (33) | 1791 (33) | 1958 (18)

9. Secondary Outcome: PF-07059013 Blood and Plasma Tmax of Part 2
Description: PF-07059013 Blood and Plasma Tmax of Part 2 was evaluated.
Time Frame: 0, 0.5, 1, 2, 4, 6, 8, 12 hours post dose on Day 1, 7, and 14.
Population: as for outcome 6
Measure: Median (Full Range); unit: hour
Arm/Group | Part 2: PF-07059013 800 mg MD With Polymer | Part 2: PF-07059013 1600 mg MD With Polymer | Part 2: PF-07059013 3000 mg MD With Polymer | Part 2: PF-07059013 4000 mg MD With Polymer
Number analyzed (Participants) | 8 | 7 | 6 | 6
hour
  Day 1 in Blood | 3.01 [2.00 to 4.08] | 4.00 [2.00 to 4.02] | 4.07 [4.03 to 6.00] | 4.02 [4.00 to 6.20]
  Day 1 in Plasma | 3.02 [1.00 to 4.08] | 4.00 [4.00 to 8.00] | 4.05 [4.00 to 8.10] | 6.00 [2.03 to 6.20]
  Day 7 in Blood: number analyzed (Participants) | 7 | 4 | 6 | 6
  Day 7 in Blood | 2.03 [2.00 to 4.00] | 4.03 [4.00 to 4.10] | 4.02 [2.00 to 4.12] | 4.03 [2.00 to 8.00]
  Day 7 in Plasma: number analyzed (Participants) | 7 | 4 | 6 | 6
  Day 7 in Plasma | 4.00 [2.00 to 12.0] | 4.07 [4.02 to 8.02] | 4.05 [2.00 to 8.00] | 5.01 [4.00 to 8.00]
  Day 14 in Blood: number analyzed (Participants) | 6 | 5 | 6 | 6
  Day 14 in Blood | 2.02 [1.00 to 12.0] | 4.00 [2.00 to 4.02] | 4.01 [2.02 to 6.00] | 4.03 [2.00 to 6.07]
  Day 14 in Plasma: number analyzed (Participants) | 6 | 5 | 6 | 6
  Day 14 in Plasma | 2.01 [2.00 to 6.02] | 4.02 [2.00 to 8.00] | 4.01 [2.00 to 8.02] | 4.03 [2.00 to 6.00]

10. Secondary Outcome: PF-07059013 Blood and Plasma Area Under the Concentration-Time Profile From Time 0 to Time Tau (AUCtau) of Part 2
Description: PF-07059013 Blood and Plasma AUCtau (the Dosing Interval, Where Tau = 24 Hours for QD Dosing) for Part 2 was evaluated.
Time Frame: 0, 0.5, 1, 2, 4, 6, 8, 12 hours post dose on Day 1, 7, and 14.
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Part 2: PF-07059013 800 mg MD With Polymer | Part 2: PF-07059013 1600 mg MD With Polymer | Part 2: PF-07059013 3000 mg MD With Polymer | Part 2: PF-07059013 4000 mg MD With Polymer
Number analyzed (Participants) | 8 | 7 | 6 | 6
ng*hr/mL
  Day 1 in Blood | 594600 (22) | 1942000 (37) | 4408000 (33) | 4884000 (34)
  Day 1 in Plasma | 5024 (15) | 8358 (24) | 16210 (18) | 18670 (37)
  Day 7 in Blood: number analyzed (Participants) | 7 | 4 | 6 | 6
  Day 7 in Blood | 1184000 (31) | 4108000 (42) | 8027000 (38) | 8666000 (18)
  Day 7 in Plasma: number analyzed (Participants) | 7 | 4 | 6 | 6
  Day 7 in Plasma | 7608 (25) | 13680 (38) | 24280 (21) | 29960 (30)
  Day 14 in Blood: number analyzed (Participants) | 6 | 5 | 6 | 6
  Day 14 in Blood | 981000 (29) | 4165000 (29) | 7730000 (21) | 9944000 (22)
  Day 14 in Plasma: number analyzed (Participants) | 6 | 5 | 6 | 6
  Day 14 in Plasma | 7568 (26) | 14330 (22) | 26500 (20) | 31640 (25)

11. Secondary Outcome: p20 and p50 (Partial Pressure of Oxygen at Which Hemoglobin is 20% or 50% Saturated With Oxygen) Change From Baseline in Part 1
Description: p20 and p50 change from baseline in Part 1 was evaluated.
Time Frame: Part 1: 0 and 8 hours post dose.
Population: The analysis population referred to all participants dosed who had at least 1 of the pharmacodynamics parameters of secondary interest.
Measure: Median (Full Range); unit: mmHg
Arm/Group | Part 1: Placebo Single Dose (SD) With Polymer | Part 1: PF-07059013 100 mg SD With Polymer | Part 1: PF-07059013 250 mg SD With Polymer | Part 1: PF-07059013 500 mg SD With Polymer | Part 1: PF-07059013 1000 mg SD With Polymer | Part 1: PF-07059013 2000 mg SD With Polymer | Part 1: PF-07059013 3000 mg SD With Polymer | Part 1: PF- 07059013 2000 mg SD Without Polymer | Part 1: PF-07059013 3000 mg SD Without Polymer
Number analyzed (Participants) | 18 | 6 | 5 | 6 | 6 | 6 | 6 | 9 | 8
mmHg
  p20 at Day 1 8H | 0.05 [-0.3 to 1.3] | 0.10 [-0.1 to 1.0] | 0.00 [-0.2 to 1.9] | -0.05 [-0.7 to 0.4] | -0.05 [-1.1 to 0.3] | -0.40 [-1.0 to -0.2] | -1.00 [-2.0 to -0.4] | -0.70 [-1.1 to -0.1] | -1.30 [-1.6 to -0.2]
  p50 at Day 1 8H | 0.50 [-0.1 to 3.3] | 0.25 [-0.2 to 1.6] | 0.20 [-0.2 to 1.6] | 0.15 [-0.9 to 1.1] | 0.50 [-1.1 to 0.9] | -0.25 [-0.7 to 0.1] | -0.45 [-1.2 to 0.1] | -0.30 [-0.9 to 0.8] | -0.45 [-1.6 to 0.4]

12. Secondary Outcome: p20 and p50 (Partial Pressure of Oxygen at Which Hemoglobin is 20% or 50% Saturated With Oxygen) Change From Baseline in Part 2
Description: p20 and p50 change from baseline in Part 2 was evaluated.
Time Frame: Part 2: 0 and 8 hours post dose on Day 1, 7 and 14, and on Day 2, 15, 18.
Population: as for outcome 11
Measure: Median (Full Range); unit: mmHg
Arm/Group | Part 2: Placebo Multiple Doses (MD) With Polymer | Part 2: PF-07059013 800 mg MD With Polymer | Part 2: PF-07059013 1600 mg MD With Polymer | Part 2: PF-07059013 3000 mg MD With Polymer | Part 2: PF-07059013 4000 mg MD With Polymer
Number analyzed (Participants) | 8 | 8 | 7 | 6 | 6
mmHg
  p20 at Day 1 2H | 0.10 [-0.6 to 0.6] | -0.30 [-1.4 to 0.2] | -0.90 [-1.1 to -0.4] | -1.25 [-2.9 to -0.4] | -2.00 [-3.8 to -0.2]
  p20 at Day 2: number analyzed (Participants) | 8 | 8 | 7 | 6 | 2
  p20 at Day 2 | 0.30 [-1.5 to 1.5] | 0.55 [-2.1 to 0.8] | -1.00 [-1.6 to 0.1] | -0.45 [-1.2 to 0.9] | -2.10 [-2.4 to -1.8]
  p20 at Day 7 0H: number analyzed (Participants) | 7 | 4 | 5 | 5 | 6
  p20 at Day 7 0H | 0.70 [-1.7 to 1.0] | -0.65 [-2.6 to 0.2] | 0.00 [-0.3 to 0.8] | -1.60 [-3.0 to 2.4] | -1.05 [-2.3 to 0.5]
  p20 at Day 7 2H: number analyzed (Participants) | 7 | 4 | 5 | 5 | 6
  p20 at Day 7 2H | 0.30 [-1.5 to 1.3] | -1.20 [-2.9 to -0.4] | -0.70 [-1.2 to -0.1] | -3.60 [-6.6 to 1.0] | -3.05 [-9.4 to 0.0]
  p20 at Day 14 0H: number analyzed (Participants) | 8 | 7 | 5 | 5 | 6
  p20 at Day 14 0H | 0.35 [-1.2 to 1.9] | 0.40 [-2.1 to 0.8] | 0.00 [-0.6 to 2.4] | -2.70 [-4.1 to -0.1] | -2.20 [-4.1 to 1.6]
  p20 at Day 14 2H: number analyzed (Participants) | 8 | 6 | 5 | 5 | 6
  p20 at Day 14 2H | 0.40 [-1.0 to 2.2] | -0.05 [-2.3 to 0.6] | -0.20 [-1.3 to 1.8] | -5.20 [-11.1 to -0.4] | -8.05 [-12.0 to 0.0]
  p20 at Day 14 24H: number analyzed (Participants) | 6 | 7 | 5 | 6 | 4
  p20 at Day 14 24H | -0.65 [-1.7 to 1.3] | 0.50 [-2.1 to 1.5] | 0.20 [-2.4 to 2.0] | -1.40 [-3.7 to 2.0] | -1.35 [-2.4 to 1.6]
  p20 at Day 14 96H: number analyzed (Participants) | 3 | 0 | 3 | 4 | 4
  p20 at Day 14 96H | -0.10 [-1.6 to 0.2] |  | 1.70 [-0.1 to 2.4] | 0.15 [-0.7 to 0.8] | 1.40 [0.8 to 3.8]
  p50 at Day 1 2H | 0.30 [-0.7 to 1.1] | 0.00 [-0.4 to 1.2] | -0.40 [-0.8 to 0.1] | -0.35 [-1.3 to 0.0] | -0.95 [-2.2 to 0.4]
  p50 at Day 2: number analyzed (Participants) | 8 | 8 | 7 | 6 | 2
  p50 at Day 2 | 0.85 [-2.0 to 2.3] | 1.00 [-4.1 to 1.5] | -0.40 [-1.0 to 0.6] | 0.25 [-0.6 to 1.1] | -1.45 [-2.0 to -0.9]
  p50 at Day 7 0H: number analyzed (Participants) | 7 | 4 | 5 | 5 | 6
  p50 at Day 7 0H | 0.60 [-3.2 to 2.2] | -1.30 [-5.6 to 1.4] | 0.70 [0.1 to 1.8] | -0.30 [-1.9 to 4.7] | 0.10 [-0.8 to 1.6]
  p50 at Day 7 2H: number analyzed (Participants) | 7 | 4 | 5 | 5 | 6
  p50 at Day 7 2H | 0.80 [-2.8 to 2.4] | -1.30 [-5.4 to 1.0] | 0.70 [-0.3 to 1.6] | -2.20 [-2.6 to 2.9] | -0.60 [-4.3 to 0.6]
  p50 at Day 14 0H: number analyzed (Participants) | 8 | 7 | 5 | 5 | 6
  p50 at Day 14 0H | 0.60 [-1.9 to 1.7] | 0.70 [-4.3 to 1.6] | 1.40 [-0.3 to 4.1] | -2.00 [-3.3 to -0.1] | -0.70 [-2.1 to 1.9]
  p50 at Day 14 2H: number analyzed (Participants) | 8 | 6 | 5 | 5 | 6
  p50 at Day 14 2H | 0.75 [-1.1 to 2.2] | 1.05 [-4.3 to 2.2] | 1.00 [-0.6 to 3.6] | -3.50 [-6.3 to -0.2] | -2.80 [-6.9 to 0.8]
  p50 at Day 14 24H: number analyzed (Participants) | 6 | 7 | 5 | 6 | 4
  p50 at Day 14 24H | -0.85 [-2.2 to 2.3] | 1.30 [-4.0 to 2.7] | 1.10 [-2.3 to 3.5] | -0.50 [-3.2 to 3.5] | 0.45 [-0.9 to 2.6]
  p50 at Day 14 96H: number analyzed (Participants) | 3 | 0 | 3 | 4 | 4
  p50 at Day 14 96H | -0.70 [-2.7 to 0.9] |  | 2.70 [1.0 to 3.2] | 0.15 [-0.4 to 1.4] | 2.90 [2.1 to 4.9]

ADVERSE EVENTS:
Time Frame: Baseline up to Follow-Up (15 weeks in Part 1 and Part 3, and 10 weeks in Part 2).
Arm/Group | Part 1: Placebo Single Dose (SD) With Polymer | Part 1: PF-07059013 100 mg SD With Polymer | Part 1: PF-07059013 250 mg SD With Polymer | Part 1: PF-07059013 500 mg SD With Polymer | Part 1: PF-07059013 1000 mg SD With Polymer | Part 1: PF-07059013 2000 mg SD With Polymer | Part 1: PF-07059013 3000 mg SD With Polymer | Part 1: PF- 07059013 2000 mg SD Without Polymer | Part 1: PF-07059013 3000 mg SD Without Polymer | Part 2: Placebo Multiple Doses (MD) With Polymer | Part 2: PF-07059013 800 mg MD With Polymer | Part 2: PF-07059013 1600 mg MD With Polymer | Part 2: PF-07059013 3000 mg MD With Polymer | Part 2: PF-07059013 4000 mg MD With Polymer | Part 3: Suspension Fasted Polymer (Small Particle Size) | Part 3: Tablet Fasted Without Polymer | Part 3: Suspension Fed Polymer (Small Particle Size)
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/6 | 0/5 | 0/6 | 0/6 | 0/6 | 0/6 | 0/9 | 0/8 | 0/8 | 0/8 | 0/7 | 0/6 | 0/6 | 0/3 | 0/4 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/6 | 0/5 | 0/6 | 0/6 | 0/6 | 0/6 | 0/9 | 0/8 | 0/8 | 0/8 | 0/7 | 0/6 | 0/6 | 0/3 | 0/4 | 0/1
Other Adverse Events (participants affected / at risk) | 3/18 | 2/6 | 2/5 | 0/6 | 1/6 | 0/6 | 4/6 | 2/9 | 4/8 | 4/8 | 7/8 | 7/7 | 4/6 | 5/6 | 3/3 | 2/4 | 0/1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Placebo Single Dose (SD) With Polymer (N=18) | Part 1: PF-07059013 100 mg SD With Polymer (N=6) | Part 1: PF-07059013 250 mg SD With Polymer (N=5) | Part 1: PF-07059013 500 mg SD With Polymer (N=6) | Part 1: PF-07059013 1000 mg SD With Polymer (N=6) | Part 1: PF-07059013 2000 mg SD With Polymer (N=6) | Part 1: PF-07059013 3000 mg SD With Polymer (N=6) | Part 1: PF- 07059013 2000 mg SD Without Polymer (N=9) | Part 1: PF-07059013 3000 mg SD Without Polymer (N=8) | Part 2: Placebo Multiple Doses (MD) With Polymer (N=8) | Part 2: PF-07059013 800 mg MD With Polymer (N=8) | Part 2: PF-07059013 1600 mg MD With Polymer (N=7) | Part 2: PF-07059013 3000 mg MD With Polymer (N=6) | Part 2: PF-07059013 4000 mg MD With Polymer (N=6) | Part 3: Suspension Fasted Polymer (Small Particle Size) (N=3) | Part 3: Tablet Fasted Without Polymer (N=4) | Part 3: Suspension Fed Polymer (Small Particle Size) (N=1)
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 2 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 0
Restless legs syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Application Site Pruritus (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Puncture Site Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thermal Burn (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
SARS-CoV-2 Test Positive (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nocturia (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Polyuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dry Skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Orthostatic Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 1 | 0 | 0 | 0
Conjunctival Hyperaemia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ocular Hyperaemia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Photophobia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal Discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abnormal faeces (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Anal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Faeces Discoloured (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chest Discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chest Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Burn Oesophageal (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Joint Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Limb Discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dizziness Postural (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Head Discomfort (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Dry Throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0
Hot Flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ear Pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tongue Haematoma (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
After the completion of the Part 1 and Part 2, due to failure to demonstrate sufficient pharmacologic effect in relation to the study PK and pharmacodynamic (PD) objectives in healthy participants as defined in the study protocol, the study was terminated prematurely. The decision to terminate the study was made while Part 3 was in progress (5 participants enrolled).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2020-07-24): https://cdn.clinicaltrials.gov/large-docs/24/NCT04323124/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-28): https://cdn.clinicaltrials.gov/large-docs/24/NCT04323124/SAP_001.pdf